CLINICAL TRIAL: NCT02864589
Title: Internet-based Behaviour Therapy for Tourette's Disorder and Chronic Tic Disorder: A Feasibility Study
Brief Title: Internet-based Behaviour Therapy for Tourette's Disorder and Chronic Tic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, David Mataix-Cols, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/938-31/4
Record Dates: First submitted 2016-08-09; First posted 2016-08-12 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Tourette's Disorder; Persistent (Chronic) Motor or Vocal Tic Disorder
Keywords: Tourette, Tic, Tics
MeSH Terms: conditions — Tourette Syndrome; Bronchiolitis Obliterans Syndrome; Tic Disorders; Tics | interventions — Hormone Replacement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- I-HRT (Experimental): Internet-delivered habit reversal training
  Interventions: Behavioral: Internet-delivered habit reversal training
- I-ERP (Experimental): Internet-delivered exposure and response prevention
  Interventions: Behavioral: Internet-delivered exposure and response prevention

INTERVENTIONS:
Behavioral: Internet-delivered habit reversal training — The I-HRT group will receive a 10-week therapist-guided, parent-assisted, Internet-delivered behavioural treatment. The treatment is based on existing literature on habit reversal training (i.e. Woods, D.W. (2008). Managing Tourette syndrome: A behavioral intervention for children and adults therapist guide. OUP, USA.) with added interactive features as videos and illustrations. In short, the participants practice to become more aware of their tics and inhibit them by performing competing responses (movements). The treatment is therapist guided: the participants have regular (up to 5 days a week) contact with a personally assigned therapist via written text in the platform and occasionally via the telephone. The children and parents have separate logins and access partly different content.
  Other Names: HRT, HR
  Arms: I-HRT
Behavioral: Internet-delivered exposure and response prevention — The I-ERP group receives a 10-week therapist-guided, parent-assisted, Internet-delivered behavioural treatment. The treatment is based on existing literature on exposure and response prevention (i.e. Verdellen, C. et al. (2011). Tics: Therapist manual & workbook for children. Boom, Amsterd.) with added interactive features as videos and illustrations. In short, the participants practice to suppress their tics for longer and longer times, at the same time as premonitory urges are intentionally provoked. The treatment is therapist-guided: the children and parents have regular (up to 5 days a week) contact with a personally assigned therapist via written text in the platform and occasionally via the telephone. The children and parents have separate logins and access partly different content.
  Other Names: ERP
  Arms: I-ERP

SUMMARY:
The purpose of this study is to evaluate the feasibility and acceptability of two different modalities of therapist-guided Internet-delivered behaviour therapy (IBT) for children and adolescents (7-17 years) with Tourette's Disorder (TD) or Persistent (Chronic) Motor or Vocal Tic Disorder (PTD).

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the feasibility and acceptability of two different modalities of therapist-guided Internet-delivered behaviour therapy (IBT) for children and adolescents (7-17 years) with Tourette's Disorder (TD) or Persistent (Chronic) Motor or Vocal Tic Disorder (PTD). The two modalities of IBT are habit reversal training (HRT) and exposure and response prevention (ERP). Secondary objectives are to evaluate whether IBT can decrease tic frequency and tic-related impairment, and, as both HRT and ERP have been proven efficacious in treating TD/PTD face-to-face, are any of the two treatments better suited to be delivered via the internet?

The design of the study is a randomized-controlled trial with 20 participants. Participants will be stratified by ADHD/ADD status.

The treatment duration is 10 weeks.

Feasibility and acceptability will be assumed if:

* The two treatments can be successfully adapted to a therapist guided internet-delivered format (technical feasibility)
* Patients/parents are willing to try the offered treatment modalities
* Participants complete the active parts of the treatment
* Referrers are open to the idea of internet-delivered treatment for TD or PTD
* We can recruit sufficient numbers of patients for a fully powered efficacy trial

Regarding the secondary objective, the primary outcome is tic severity measured by the Yale Global Tic Severity Scale (YGTSS). Participants will be assessed directly after treatment (post), and at 3, 6 and 12 months after treatment. Assessments at post-treatment and 3 month follow up will be performed by assessors blinded to the treatment condition. After 3 months, we will naturalistically follow up patients up to 12 months after the end of treatment. Data collection will finish 12 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill DSM-5 diagnostic criteria for Tourette's Disorder or Persistent (Chronic) Motor or Vocal Tic Disorder (PTD).
* >15 (TD) or >10 (PTD) on Yale Global Tic Severity Scale (Impairment not included).
* Both child and parent are able to read and communicate in Swedish.
* Regular access to a computer and the Internet.
* Parent availability to support their child throughout the treatment.

Exclusion Criteria:

* Acute psychiatric problems such as severe depression, suicidal risk, substance abuse or another psychiatric disorder that could interfere with treatment.
* Lifetime history of global learning disability, pervasive developmental disorder, psychosis, bipolar disorder or organic brain disorder.
* Severe tics causing immediate risk to the patients or others and requiring urgent medical attention.
* Previous behavioural therapy (HRT or ERP), minimum 8 sessions with qualified therapist, within the last 12 months prior to assessment.
* Simultaneous psychological treatment for tic disorder.
* Initiation or adjustment of any psychotropic medication for tics within the last 6 weeks prior to assessment.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2016-08; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Yale Global Tic Severity Scale (YGTSS) | Week 0; week 10; 3 months follow up; 6 months follow up; 12 months follow up
  Change in tic severity (motor and/or vocal tics) from week 0 (pre treatment) to week 10 (post treatment), 3 months follow up (after post treatment), 6 months follow up and 12 months follow up.

SECONDARY OUTCOMES:
Clinical Global Impression - Severity (CGI-S) | Week 0; week 10; 3 months follow up; 6 months follow up; 12 months follow up
Clinical Global Impression - Improvement (CGI-I) | Week 10; 3 months follow up; 6 months follow up; 12 months follow up
Children's Global Assessment Scale (C-GAS) | Week 0; week 10; 3 months follow up; 6 months follow up; 12 months follow up
Parent Tic Questionnaire (PTQ) | Week 0; week 5; week 10; 3 months follow up; 6 months follow up; 12 months follow up
Premonitory urge for Tics Scale (PUTS) | Week 0; week 5; week 10; 3 months follow up; 6 months follow up; 12 months follow up
Gilles de la Tourette Syndrome Quality of Life Scale (GTS-QOL). | Week 0; week 10; 3 months follow up; 6 months follow up; 12 months follow up
Obsessive-Compulsive Inventory - Child version (OCI-CV). | Week 0; week 10; 3 months follow up; 6 months follow up; 12 months follow up
Children's Depression Inventory - Short version (CDI-S), with additional suicidality item | Week 0; week 5; week 10; 3 months follow up; 6 months follow up; 12 months follow up
Mood and Feeling Questionnaire - Short version (MFQ) | Week 0; week 5; week 10; 3 months follow up; 6 months follow up; 12 months follow up
Education, Work and Social Adjustment Scale - Child version (EWSAS-C) | Week 0; week 10; 3 months follow up; 6 months follow up; 12 months follow up
Education, Work and Social Adjustment Scale - Parent version (EWSAS-P) | Week 0; week 10; 3 months follow up; 6 months follow up; 12 months follow up
Treatment credibility scale | Week 3
Treatment satisfaction scale | Week 10
Safety Monitoring Uniform Report Form (SMURF) | Week 5; week 10
Internet Intervention Patient Adherence Scale (iiPAS) | Week 5; week 10
Parental strategy scale | Week 10

CONTACTS AND LOCATIONS:
Overall Officials: David Mataix-Cols, Professor, Principal Investigator — Karolinska Institutet, Department of Clinical Neuroscience
Locations (1):
- BUP CPF, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Andren P, Aspvall K, Fernandez de la Cruz L, Wiktor P, Romano S, Andersson E, Murphy T, Isomura K, Serlachius E, Mataix-Cols D. Therapist-guided and parent-guided internet-delivered behaviour therapy for paediatric Tourette's disorder: a pilot randomised controlled trial with long-term follow-up. BMJ Open. 2019 Feb 15;9(2):e024685. doi: 10.1136/bmjopen-2018-024685. PMID 30772854